CLINICAL TRIAL: NCT00486148
Title: Randomized, Double Blind Study to Evaluate the Safety and Efficacy of an Infant Formula Supplemented With Galacto-oligosaccharides (GOS) in Healthy, Full Term Infants
Brief Title: Safety and Efficacy of an Infant Formula Supplemented With Galacto-oligosaccharides (GOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinz Italia SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLA-1-GOS-05
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Nutritional Safety
Keywords: Formula; Feeding; Healthy; Full; Term; Infants
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- group "S" (No Intervention): Breast milk
- group "A" (No Intervention): Control Infant formula
- group "B" (Experimental): Infant formula supplemented with 0.4 g/100 ml of oligosaccharides
  Interventions: Other: Infant formula (with GOS)

INTERVENTIONS:
Other: Infant formula (with GOS) — Infant formula supplemented with 0.4 g/100 ml of galacto-oligosaccharides
  Arms: group "B"

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an infant formula supplemented with a "prebiotic" component (GOS) in improving the gut microflora balance, mimicking that of breast-fed infants.

DETAILED DESCRIPTION:
Oligosaccharides are one of the major breast milk components. They are not digested and reach the colon where they're used by selected groups of microflora positive bacteria, specifically bifidobacteria and lactobacilli.

Therefore, oligosaccharides have prebiotic effects accountable for health benefits in infants.

Over the last years the supplementation of infant formulae has been studied to mimic breast milk prebiotic functions enhancing gut microflora growth similar to that of breast fed infants.

However further scientific data are necessary to support the efficacy of the supplementation of oligosaccharide in infant formulae.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants of both sexes, born at term with natural labor or cesarean birth
2. Single birth
3. Infant born between 37th - 42th gestation week (included)
4. Infant with birth weight ≥ 2500 g
5. APGAR score after 5 minutes of life > 7
6. Infant born from parents of Caucasian race
7. Exclusive breast feeding or formula feeding within 15 days from birth.
8. Consensus form signed by both parents or by the legal tutor properly informed of the study.
9. Parents able to understand the protocol requirements and to fill out the infants Diary.

Exclusion Criteria:

1. Infant with inborn malformation and with hereditary and/or chronic and/or inborn diseases requiring hospital care superior to 7 days.
2. Diseases jeopardizing intrauterine growth.
3. Infant born from mother suffering from dismetabolic and/or chronic diseases.
4. Unknown father
5. Infant with parents who might not report at hospital controls or not follow the protocol.
6. Infant already enrolled or selected for another clinical trial.

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2006-02; Primary Completion 2011-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The nutritional safety through anthropometric controls. Adverse events: diarrhea, crying, gaseous colics, regurgitation, vomit, skin rashes, fever. | Anthropometric controls at birth, on enrolment, after 1, 2, 3, 4 months of life and just before starting weaning. Adverse events daily.

SECONDARY OUTCOMES:
The prebiotic effect through the control of the feces consistency and frequency, the incidence of gaseous colics and microbiological analyses of the fecal samples. | Feces consistency and frequency, and incidence of gaseous colics, microbiological analyses of the fecal samples on enrolment and after 1 and 2 months of life.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Agostoni, Prof, Principal Investigator — Azienda Ospedaliera San Paolo; Gian Vincenzo Zuccotti, Prof, Principal Investigator — Azienda Ospedaliera "Luigi Sacco"; Giacomo Biasucci, Dr, Principal Investigator — Ospedale Civile "G. da Saliceto"; Fabio Alberto Podestà, Dr, Principal Investigator — Ospedale San Carlo Borromeo; Amilcare Rottoli, Dr, Principal Investigator — "Casa Pia Ospitaliera Uboldo" - Ospedale "Santa Maria delle Stelle"; Cino Galluzzo, Dr, Principal Investigator — Ospedale "Sacra Famiglia del Fatebenefratelli"
Locations (7):
- Italy (7):
  - "Casa Pia Ospitaliera Uboldo" Unità Operativa di Pediatria e Neonatologia, Cernusco Sul Naviglio (Milan)
  - Ospedale "Sacra Famiglia del Fatebenefratelli" Unità Operativa di Pediatria e Neonatologia, Erba (Como)
  - Ospedale "Santa Maria delle Stelle" Unità Operativa di Pediatria e Neonatologia, Melzo (MI)
  - Azienda ospedaliera "San Paolo", Dipartimento di Pediatria, Milan
  - Ospedale "San Carlo Borromeo" Unità Operativa di Pediatria, Milan
  - Azienda Ospedaliera "Luigi Sacco" Unità Operativa di Pediatria, Milan
  - Ospedale Civile "G. da Saliceto" Unità Operativa di Pediatria, Piacenza

REFERENCES:
- [Background] Mountzouris KC, McCartney AL, Gibson GR. Intestinal microflora of human infants and current trends for its nutritional modulation. Br J Nutr. 2002 May;87(5):405-20. doi: 10.1079/BJNBJN2002563. PMID 12010580
- [Background] Agostoni C, Axelsson I, Goulet O, Koletzko B, Michaelsen KF, Puntis JW, Rigo J, Shamir R, Szajewska H, Turck D; ESPGHAN Committee on Nutrition. Prebiotic oligosaccharides in dietetic products for infants: a commentary by the ESPGHAN Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2004 Nov;39(5):465-73. doi: 10.1097/00005176-200411000-00003. PMID 15572882
- [Background] Gibson GR, Roberfroid MB. Dietary modulation of the human colonic microbiota: introducing the concept of prebiotics. J Nutr. 1995 Jun;125(6):1401-12. doi: 10.1093/jn/125.6.1401. PMID 7782892
- [Background] Macfarlane GT, Cummings JH. Probiotics and prebiotics: can regulating the activities of intestinal bacteria benefit health? BMJ. 1999 Apr 10;318(7189):999-1003. doi: 10.1136/bmj.318.7189.999. No abstract available. PMID 10195977
- [Background] Moro G, Minoli I, Mosca M, Fanaro S, Jelinek J, Stahl B, Boehm G. Dosage-related bifidogenic effects of galacto- and fructooligosaccharides in formula-fed term infants. J Pediatr Gastroenterol Nutr. 2002 Mar;34(3):291-5. doi: 10.1097/00005176-200203000-00014. PMID 11964956
- [Background] Boehm G, Lidestri M, Casetta P, Jelinek J, Negretti F, Stahl B, Marini A. Supplementation of a bovine milk formula with an oligosaccharide mixture increases counts of faecal bifidobacteria in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2002 May;86(3):F178-81. doi: 10.1136/fn.86.3.f178. PMID 11978748
- [Background] Schmelzle H, Wirth S, Skopnik H, Radke M, Knol J, Bockler HM, Bronstrup A, Wells J, Fusch C. Randomized double-blind study of the nutritional efficacy and bifidogenicity of a new infant formula containing partially hydrolyzed protein, a high beta-palmitic acid level, and nondigestible oligosaccharides. J Pediatr Gastroenterol Nutr. 2003 Mar;36(3):343-51. doi: 10.1097/00005176-200303000-00008. PMID 12604972
- [Background] Long SS, Swenson RM. Development of anaerobic fecal flora in healthy newborn infants. J Pediatr. 1977 Aug;91(2):298-301. doi: 10.1016/s0022-3476(77)80836-6. PMID 874690
- [Background] Rotimi VO, Duerden BI. The development of the bacterial flora in normal neonates. J Med Microbiol. 1981 Feb;14(1):51-62. doi: 10.1099/00222615-14-1-51. PMID 7463467
- [Background] Orrhage K, Nord CE. Factors controlling the bacterial colonization of the intestine in breastfed infants. Acta Paediatr Suppl. 1999 Aug;88(430):47-57. doi: 10.1111/j.1651-2227.1999.tb01300.x. PMID 10569223
- [Background] Benno Y, Sawada K, Mitsuoka T. The intestinal microflora of infants: composition of fecal flora in breast-fed and bottle-fed infants. Microbiol Immunol. 1984;28(9):975-86. doi: 10.1111/j.1348-0421.1984.tb00754.x. PMID 6513816
- [Background] Lundequist B, Nord CE, Winberg J. The composition of the faecal microflora in breastfed and bottle fed infants from birth to eight weeks. Acta Paediatr Scand. 1985 Jan;74(1):45-51. doi: 10.1111/j.1651-2227.1985.tb10919.x. PMID 3984727
- [Background] Howie PW. Protective effect of breastfeeding against infection in the first and second six months of life. Adv Exp Med Biol. 2002;503:141-7. doi: 10.1007/978-1-4615-0559-4_16. No abstract available. PMID 12026013
- [Background] Heine W, Mohr C, Wutzke KD. Host-microflora correlations in infant nutrition. Prog Food Nutr Sci. 1992;16(2):181-97. PMID 1496120
- [Background] Kunz C, Rodriguez-Palmero M, Koletzko B, Jensen R. Nutritional and biochemical properties of human milk, Part I: General aspects, proteins, and carbohydrates. Clin Perinatol. 1999 Jun;26(2):307-33. PMID 10394490
- [Background] Kunz C, Rudloff S, Baier W, Klein N, Strobel S. Oligosaccharides in human milk: structural, functional, and metabolic aspects. Annu Rev Nutr. 2000;20:699-722. doi: 10.1146/annurev.nutr.20.1.699. PMID 10940350
- [Background] Engfer MB, Stahl B, Finke B, Sawatzki G, Daniel H. Human milk oligosaccharides are resistant to enzymatic hydrolysis in the upper gastrointestinal tract. Am J Clin Nutr. 2000 Jun;71(6):1589-96. doi: 10.1093/ajcn/71.6.1589. PMID 10837303
- [Background] Erney RM, Malone WT, Skelding MB, Marcon AA, Kleman-Leyer KM, O'Ryan ML, Ruiz-Palacios G, Hilty MD, Pickering LK, Prieto PA. Variability of human milk neutral oligosaccharides in a diverse population. J Pediatr Gastroenterol Nutr. 2000 Feb;30(2):181-92. doi: 10.1097/00005176-200002000-00016. PMID 10697138
- [Background] Giovannini M, Riva E, Banderali G, Scaglioni S, Veehof SH, Sala M, Radaelli G, Agostoni C. Feeding practices of infants through the first year of life in Italy. Acta Paediatr. 2004 Apr;93(4):492-7. doi: 10.1080/08035250410025591. PMID 15188977
- [Background] Howie PW, Forsyth JS, Ogston SA, Clark A, Florey CD. Protective effect of breast feeding against infection. BMJ. 1990 Jan 6;300(6716):11-6. doi: 10.1136/bmj.300.6716.11. PMID 2105113
- [Background] Kramer MS, Kakuma R. Optimal duration of exclusive breastfeeding. Cochrane Database Syst Rev. 2002;(1):CD003517. doi: 10.1002/14651858.CD003517. PMID 11869667